CLINICAL TRIAL: NCT00806000
Title: Prevalence of Exercise-Induced Asthma in Select Cohorts of College Athletes
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jonathan Parsons, M.D., Ohio State University
Other Study IDs: 2008H0094
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
Keywords: Prevalence of Exercised induced asthma in athletes
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Athletes

SUMMARY:
This study is investigating how commonly exercise-induced asthma happens in athletes and the best way to diagnose exercise-induced asthma. Exercise-induced asthma describes narrowing of the airways in the lungs that occurs in certain people when they exercise. This can cause shortness of breath, cough, and fatigue during exercise and can impair athletic performance. Exercise-induced asthma can be difficult to diagnose. This is a research study, because the investigators are examining the best way to document a diagnosis of exercise-induced asthma. The investigators are also interested in examining why exercise-induced asthma may occur.

DETAILED DESCRIPTION:
prospective, cohort study of the prevalence of asthma in select athletic teams at a large, collegiate athletic program as documented by self-report versus lung function testing. Athletes from men's and women's ice hockey, soccer, and lacrosse will be studied. Each athlete will indicate via self-report on questionnaires whether they have asthma, and then subsequently will be tested utilizing specialized lung function testing. These teams were chosen, because it will allow for gender-matching across teams and they had subjectively reported asthma prevalence rates based on prior pilot data.

Inclusion Criteria:

1. Varsity athlete on athletic team of interest here at The Ohio State University
2. 18 years of age or older
3. No short-acting bronchodilator use for 6 hours prior to testing
4. No long-acting bronchodilator use for 36 hours prior to testing
5. No inhaled corticosteroids or leukotriene modifiers for 72 hours prior to testing
6. Non-smoker for 6 months or longer
7. Less than 10 pack year (number of packs per day (x) years of smoking=pack years) smoking history, as smoking causes chronic changes in the profile of inflammatory cells of lungs and also makes airways more likely to spasm. This is true even for non-smokers.

Exclusion criteria:

1. pregnancy
2. recent upper respiratory tract infection (within 2 weeks of study enrollment)
3. Objective evidence of severe lung impairment on pulmonary testing performed at the beginning of the study.
4. Participation in another interventional research trial
5. Unable to provide consent
6. Asthma exacerbation within the last 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Varsity athlete on athletic team of interest here at The Ohio State University
* 18 years of age or older
* No short-acting bronchodilator use for 6 hours prior to testing
* No long-acting bronchodilator use for 36 hours prior to testing
* No inhaled corticosteroids or leukotriene modifiers for 72 hours prior to testing
* Non-smoker for 6 months or longer
* Less than 10 pack year (number of packs per day (x) years of smoking=pack years) smoking history, as smoking causes chronic changes in the profile of inflammatory cells of lungs and also makes airways more likely to spasm. This is true even for non-smokers

Exclusion Criteria:

* pregnancy
* recent upper respiratory tract infection (within 2 weeks of study enrollment)
* Objective evidence of severe lung impairment on pulmonary testing performed at the beginning of the study.
* Participation in another interventional research trial
* Unable to provide consent
* Asthma exacerbation within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: select athletic teams including men and women's ice hockey, soccer, and lacross
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

SECONDARY OUTCOMES:
To identify characteristics of athletes that may be associated with increased relative risk for asthma To identify characteristics of athletes that may be associated with increased relative risk for asthma. To identify characteristics of athletes tha | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Parsons, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States